CLINICAL TRIAL: NCT06941428
Title: Systematic Redesign of Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) to Enhance Usability, Engagement, Appropriateness, and Impact in Schools
Brief Title: Systematic Redesign of Trauma-Focused Cognitive Behavioral Therapy (TF-CBT)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Aaron Lyon, Professor, Department of Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00019451; P50MH115837 (NIH)
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Trauma, Psychological; Trauma and Stressor Related Disorders
Keywords: School Mental Health; Trauma-Focused Cognitive Behavioral Therapy
MeSH Terms: conditions — Psychological Trauma; Trauma and Stressor Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) (Active Comparator): Participants in this arm will receive TF-CBT gold-standard training and 6 months of follow-up consultation will be delivered by a certified trainer.
  Interventions: Behavioral: Trauma-Focused Cognitive Behavioral Therapy (TF-CBT)
- School-Adapted TF-CBT (S-TF) (Experimental): Participants in this arm will receive S-TF training and consultation procedures will align with those for TF-CBT to ensure comparable training/consultation dose.
  Interventions: Behavioral: School-Adapted TF-CBT (S-TF)

INTERVENTIONS:
Behavioral: Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) — TF-CBT is a cognitive-behavioral individual intervention for children aged 3 to 18 years with trauma exposure and related mental health sequelae.TF-CBT core components include psychoeducation, relaxation skills, affective regulation skills, cognitive coping skills, construction of a trauma narrative to facilitate imaginal exposure and cognitive processing of the traumatic events, and in vivo exposure to trauma reminders. TF-CBT is hypothesized to operate on specific mechanisms that influence improvements in clinical outcomes.
  Arms: Trauma-Focused Cognitive Behavioral Therapy (TF-CBT)
Behavioral: School-Adapted TF-CBT (S-TF) — S-TF is a version of Trauma-Focused Cognitive Behavioral Therapy modified for delivery by providers in the education sector. Although modifications will be determined by Study 1 activities, we anticipate that S-TF might modify treatment pacing, session length, or content sequencing. Regardless, the core functions of TF-CBT will be retained in the S-TF redesign.
  Arms: School-Adapted TF-CBT (S-TF)

SUMMARY:
Trauma-focused cognitive behavior therapy (TF-CBT) has the strongest evidence of any clinical intervention for youth trauma but is rarely adopted in the education sector - the most common setting for youth mental healthcare. Use of TF-CBT in schools is limited by (1) problems with its usability (e.g., rigid structures, complicated patient identification workflows) and (2) provider perceptions that some core elements (e.g., exposure) are not contextually appropriate for schools; both of which hinder provider and student engagement with TF-CBT. Our preliminary studies identified that TF-CBT demonstrates "below average" usability, suggesting that many providers are likely to experience it as excessively onerous (e.g., due to lengthy sessions, low caregiver engagement). Without a systematic process for redesign, treatment adaptations made to improve intervention-setting fit can be reactive and risk omitting their core elements or functions. Locally driven, user focused redesign of TF-CBT for schools that maintains its core functions can enhance the accessibility and impact of evidence-based trauma treatment for youth. In light of the need for usable, contextually appropriate, and engaging interventions for youth trauma, the current project will iteratively adapt TF-CBT for use by school-based providers (e.g., school counselors, school social workers) via the University of Washington ALACRITY Center's (UWAC) Discover, Design/Build, Test (DDBT) approach and methods drawn from the field of human-centered design.

DETAILED DESCRIPTION:
The investigators will compare DDBT mechanisms (usability, engagement, appropriateness) and implementation outcomes (adoption, fidelity, adaptation, reach) for local school-adapted TF-CBT (S-TF) versus original TF-CBT (TF-CBT). Although the content of the intervention will be redesigned, basic training format and implementation structures (e.g., online training, live workshop, role plays, consultation) will be held constant across conditions. The investigators hypothesize:

H-1: S-TF will demonstrate greater usability, engagement, and appropriateness than TF-CBT.

H-2: S-TF will demonstrate greater adoption, fidelity, reach, degree of implementation, and fewer reactive adaptations, than TF-CBT.

The investigators will also evaluate the potential impact of S-TF versus TF-CBT for students experiencing elevated trauma symptoms on TF-CBT mechanisms (trauma-related cognitions, emotion regulation, behavioral avoidance) and mental health outcomes (e.g., symptoms of post-traumatic stress). The investigators hypothesize:

H-3: Across conditions, more clients will experience significant clinical improvement than will deteriorate or remain unchanged.

H-4: S-TF will demonstrate noninferiority to TF-CBT on treatment mechanisms (trauma-related cognitions, emotional regulation, and behavioral avoidance).

H-5: S-TF will demonstrate noninferiority to TF-CBT on student mental health outcomes (symptoms).

ELIGIBILITY:
INCLUSION CRITERIA

Discover, Design/Build Phase:

* Providers. Providers will be included if they (a) deliver mental health treatment on school grounds; (b) English speaking.
* Students. Youth participants will meet eligibility criteria for this study, including (a) be within the TF-CBT developmental range, ages 7-19; (b) are receiving, or have previously received, school mental health services; and (c) are English speaking.

Test Phase:

* Providers. Providers will be included if they (a) deliver mental health treatment on school grounds; (b) have not previously received formal training in TF-CBT; and (c) are English speaking
* Students. Youth participants will meet eligibility criteria for this study, including (a) be within the TF-CBT developmental range, ages 7-19; (b) have traumatic event exposure (e.g., exposure to violence); (c) demonstrate significant post-traumatic stress symptoms (have a trauma history as defined as a score >31 on the Child PTSD Symptoms Scale for DSM-V [CPSS-V]); and (d) are English speaking.

EXCLUSION CRITERIA

Discover, Design/Build Phase:

- Students with intellectual impairments documented in education or mental health records.

Test Phase:

* Providers. Providers will be excluded if they participated in the redesign process for TF-CBT.
* Students. Students will be excluded if they (a) have intellectual impairments documented in education or mental health records and (2) are not trauma exposed.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Usability Scale (IUS) score | Baseline, 3 months, 6 months
  Usability will be evaluated with the 10-item Intervention Usability Scale (IUS), which is based closely on the well-validated SUS. Ratings are on a 1 to 5 scale and yield a total score from 0 to 100.Half the items are reverse scored; higher total scores reflect greater usability. The IUS has good inter-item consistency (a = .83) and sensitivity. Research has also demonstrated that the original version of the IUS (the SUS) function similarly, and yields similar scores, for adults and youth as young as 11 years. For youth <11, we will use an adapted lUS, modeled after an adapted version of the SUS for children as young as 7 years old and demonstrating adequate to good reliability.
Change in Participant Responsiveness Scale (PRS) score | Baseline, 3 months, 6 months
  Engagement will be measured using the Participant Responsiveness Scale (PRS), an adapted version of the 12-item Patient Responsiveness Scale tailored to be developmentally appropriate for children aged 8 and above as well as adults. The PRS measures two factors, Participation and Enthusiasm. The original Patient Responsiveness Scale has demonstrated strong reliability (a = .86) and construct validity.
Change in Intervention Appropriateness Measure (IAM) score | Baseline, 3 months, 6 months
  The Intervention Appropriateness Measure (IAM) is a rigorously developed, pragmatic instrument with strong good internal consistency (a = .87) and test-retest reliability (a = .87).
Adoption over time | End of the individual's study participation period, assessed as the study withdrawal date or 24 months post-enrollment, whichever is first
  Adoption is operationalized as the initiation of a clinician's first TF-CBT or S-TF session at any point during study participation. These data will be collected from an online Toolkit that facilitates tracking of services delivered and has been commonly used for large-scale TF-CBT implementation.
Reach over time | End of the individual's study participation period, assessed as the study withdrawal date or 24 months post-enrollment, whichever is first
  Reach will be calculated using adoption data as the percentage of clinician's caseloads receiving TF-CBT or S-TF.
Change in Child Post-Traumatic Cognitions Inventory (CPTI) score | Baseline, 3 months, 6 months
  The Child Post-Traumatic Cognitions Inventory (CPTI) is a 25-item measure for youth aged 6-18 that is applicable to a wide range of trauma experiences. Two subscales, (1) Permanent and disturbing change (in response to trauma) and (2) Fragile person in a scary world have been identified. Both subscales have high internal consistency (a = .91 and .87, respectively)and test-retest reliability (r= .78 and .72).
Change in Emotion Regulation Questionnaire-Child and Adolescent (ERQ-CA) score | Baseline, 3 months, 6 months
  The Emotion Regulation Questionnaire-Child and Adolescent (ERQ-CA) is a 10-item instrument that has demonstrated good construct validity, inter-item consistency (a = .73 - .79), and test-retest reliability (r = .69) across multiple studies for children aged 7-18 years.
Change in Posttraumatic Avoidance Behavior Questionnaire (PABQ) score | Baseline, 3 months, 6 months
  The Posttraumatic Avoidance Behavior Questionnaire (PABQ) is a 25-item self-report measuring trauma-related avoidance behavior (e.g., avoiding visual trauma reminders, being alone, intimate relationships) on a 4-point Likert scale. The PABQ has good test-retest validity (r = .87 - .78) and convergent validity with PTSD symptom severity (r= .77 - .56).
Change in Child PTSD Symptoms scale for DSM-V (CPSS-V) score | Baseline, 3 months, 6 months
  The Child PTSD Symptoms scale for DSM-V (CPSS-V) includes 20 self-report symptom items (assessed over the past month) that map onto the diagnostic criteria in DSM-5 for PTSD, items are rated 0 (not at all) to 4 (6 or more times a week/almost always) based on the frequency and severity of the reported symptom experienced. The CPSS-V has demonstrated good internal consistency (a =.92) and test-retest reliability (r= .80). A 6-item screener version of the CPSS-V is also available, which demonstrates adequate internal consistency a = .78) and test-retest reliability (r = .71, p < .001) and will be used to initially identify youth for study participation.
Change in Children Depression Inventory (CDI) score | Baseline, 3 months, 6 months
  The Children Depression Inventory (CDI) assesses cognitive, affective, and behavioral symptoms of depression during the past 2 weeks with 26 items.The CDI has good test-retest reliability and validity.
Youth Top Problems (YTP) over time | Baseline, 3 months, 6 months
  The Youth Top Problems (YTP) assessment is an assessment in which youth and caregivers are asked to list the problems they were most concerned about. Upon completion of the list, respondents are asked to assign a severity rating for each problem by answering the questions: how big of a problem is this for you?(0 = not at all to 10 = very, very much). Respondents are then asked to identify which of the problems listed: is the biggest problem right now? Which one is the most important to work on?. Then the second and third most important until 3 top problems are identified. The YTP shows excellent concurrence with standardized assessments (Kappa ranging from .78 to .91), while also adding specificity for treatment targets (41% of caregivers-, and 79% of youth-identified top problems were not identified by an item amongst elevated standardized assessment sub-scales).
Change in Quality of Life in Neurological Disorders Social Relations scale (Neuro-QOL) score | Baseline, 3 months, 6 months
  The Quality of Life in Neurological Disorders Social Relations scale (Neuro-QOL) is a widely used 8-item measure of functioning in usual social roles, activities, and responsibilities. Factor analyses and Item Response Theory analyses have ensured broad information parameters without differential item functioning by demographics. Scale scores have been validated and normed on thousands of participants in the US general and clinical inpatient and outpatient settings, presenting with a variety of problem areas. Scores provide a T score with a mean of 50 and SD of 10, aligned with a variety of norming samples. An example item stem is: In the past 7 days I am able to do all of my regular family activities. Response options are on a scale of 1 to 5 (1=never, 2=rarely, 3=sometimes, 4=often, 5=always）

SECONDARY OUTCOMES:
Therapy Process Observational Coding System (TPOCS) | Expert clinicians review audiotapes of therapy sessions for each clinician participant over a six-month period of time after initial training
  For each case, one recording will be randomly selected from each TF-CBT / S-TF treatment phase and coded for fidelity using the Therapy Process Observational Coding System (TPOCS), and the TPOCS-SeRTIF self-report measure version.
Framework for Modifications and Adaptations of Evidence-Based Intervention | End of the individual's study participation period, assessed as the study withdrawal date or 24 months post-enrollment, whichever is first
  Recorded intervention sessions will be evaluated using the coding system for the Framework for Modifications and Adaptations of Evidence-based interventions (FRAME), the leading method for evaluating the nature of intervention adaptations.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Lyon, PhD, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No